CLINICAL TRIAL: NCT01142817
Title: Metabolic and Psychological Changes Associated With Menopause Among Women With HIV
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara E. Dolan Looby, PhD, ANP-BC, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2009P-001315
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; Menopause
Keywords: HIV; Women; Menopause; Dyslipidemia; Bone Mineral Density
MeSH Terms: conditions — HIV Infections; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV Postive Women: Women living with HIV who meet study eligibility criteria
- Healthy Control Subjects: Women without HIV who meet study eligibility criteria

SUMMARY:
This study will investigate the prevalence and extent of both metabolic and psychosocial changes associated with the menopause transition over 1 year among women with HIV compared to women without HIV of similar age, weight, menstrual status, and ethnic background. It is hypothesized that HIV positive women will demonstrate increased abdominal fat, abnormal cholesterol and blood sugar levels, reduced bone density, and greater psychosocial challenges than HIV negative women during the menopause transition.

DETAILED DESCRIPTION:
Treatment with combination antiretroviral therapy (ART) has resulted in substantial improvement in survival among women living with HIV in the United States, many of whom have entered or will soon enter the menopause transition. Significant changes are seen across the menopause transition among women without HIV including increased abdominal fat and waist circumference, reduced muscle mass, and changes in lipids, glucose metabolism and bone density. HIV and potentially ART use have been associated with similar manifestations such as reduced bone density, changes in lipid and glucose metabolism, and body composition, though little is known regarding how the virus may influence or exacerbate such changes across the menopause transition. In addition to metabolic factors, menopause has been associated with changes in mood state, decreased quality of life, and presence of vasomotor symptoms among women without HIV. Psychosocial indices, such as depression and decreased quality of life are common among women with HIV, and may manifest or worsen during the menopause transition. However, research investigating the presence and acuity of these symptoms among women with HIV during menopause is limited.

ELIGIBILITY:
Inclusion Criteria:

1. Females age 45 -52.
2. Females in the perimenopausal transition characterized by the presence of abnormal menstrual function, defined as less than 3 periods in the past 3 months, 1 cycle >60 days in length in the prior 6 months, or irregular menses in 2 or more cycles within the past 6 months. Women who have been amenorrheic for >12 months will not be eligible. 3. Women with HIV must have previously documented HIV and be receiving a stable treatment regimen for > 3 months.

Exclusion Criteria:

1. Use of estrogen, combination hormone replacement therapy, oral contraceptive pills/patches, Depo Provera, glucocorticoids, testosterone, growth hormone or other anabolic steroids within the past 6 months.
2. Diabetes and current use of insulin, or medications known to affect glucose or insulin levels.
3. Positive pregnancy test or recently pregnant within the past year or lactating.
4. Presence of active cancers.
5. Current use of bisphosphonates, or a diagnosis of Paget's disease or other illnesses known to affect bone (Use of calcium and Vitamin D will be permitted).
6. Opportunistic infection within 3 months of study participation (HIV positive subjects).

   -

Ages: 45 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female subjects in the perimenopausal transition will be recruited via referral by infectious disease providers, newspaper advertisement, posted flyers, community based programs at local AIDS Service Organizations and Partners subject recruitment broadcast at Massachusetts General Hospital (MGH). The HIV negative control subjects will be recruited through advertisements, flyers, and email announcements. Both HIV positive and negative subjects will be recruited from the same neighborhoods to ensure similar demographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | baseline to 12 months
  Measurement of bone density at the toal body, lumbar spine and total hip

SECONDARY OUTCOMES:
Body Composition | baseline to 12 months
  Total body fat and abdominal fat measurement, and total lean mass measurement
Lipid Levels | baseline to 12 months
  Lipid levels include total cholesterol, low density lipoprotein, high density lipoprotein, and triglyceride levels
Glucose Metabolism | baseline to 12 months
  Includes fasting glucose and insulin levels
Depression | baseline to 12 months
  Depressive symptoms assessed by the Centers for Epidemiologic Studies Depression Scale (CES-D)
Quality of Life | baseline to 12 months
  Assessed by the Utian Quality of Life Scale
Vasomotor Symptoms | Baseline to 12 months
  Assessed by the Menopause Rating Scale, includes hot flashes, mood, sleep, genitourinary symptoms, and sexual function
Systemic Inflammation (as it relates to cardiovascular risk/body composition changes) | Baseline to 12 months
  Assessment of inflammatory biomarkers and cytokines including CRP,IL-6, TNF-α, and PAI-1, as well as adiponectin.

CONTACTS AND LOCATIONS:
Overall Officials: Sara E Looby, PhD, ANP, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Looby SE. Menopause-associated metabolic manifestations and symptomatology in HIV infection: a brief review with research implications. J Assoc Nurses AIDS Care. 2012 May-Jun;23(3):195-203. doi: 10.1016/j.jana.2011.06.008. Epub 2011 Sep 15. PMID 21924646
- [Derived] Looby SE, Shifren J, Corless I, Rope A, Pedersen MC, Joffe H, Grinspoon S. Increased hot flash severity and related interference in perimenopausal human immunodeficiency virus-infected women. Menopause. 2014 Apr;21(4):403-9. doi: 10.1097/GME.0b013e31829d4c4c. PMID 23820600